CLINICAL TRIAL: NCT03119636
Title: A Phase I/II, Open-Label Study to Assess the Safety and Efficacy of Striatum Transplantation of Human Embryonic Stem Cells-derived Neural Precursor Cells in Patients With Parkinson's Disease
Brief Title: Safety and Efficacy Study of Human ESC-derived Neural Precursor Cells in the Treatment of Parkinson's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Qi Zhou, Deputy director of Institute of zoology, Chinese academy of sciences, and vice president of medical school， University of Chinese academy of sciences, Chinese Academy of Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChineseASZQ-003
Record Dates: First submitted 2017-04-06; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2016-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NPC transplantation (Experimental): The patients will receive Levodopa combined with a regular neural precursor cell (NPC) transplantation
  Interventions: Biological: NPC transplantation; Drug: Levodopa
- HLA-matched NPC transplantation (Experimental): The patients will receive Levodopa combined with a HLA-matched neural precursor cell (NPC) transplantation
  Interventions: Biological: NPC transplantation; Drug: Levodopa
- HLA-non-matched NPC transplantation (Experimental): The patients will receive Levodopa combined with a HLA-non-matched neural precursor cell (NPC) transplantation
  Interventions: Biological: NPC transplantation; Drug: Levodopa

INTERVENTIONS:
Biological: NPC transplantation — The cells are stereotactically implanted in the striatum.
Drug: Levodopa — Levodopa is used depending on the patient's condition

SUMMARY:
This study will evaluate the safety and efficacy of intracerebral transplantation of human embryonic stem cells-derived neural precursor cells in patients with Parkinson's Disease.

DETAILED DESCRIPTION:
This study is a Phase I/II, open-label, non randomized clinical trial. The study will enroll 50 patients for cell injection, administering a single dose of neural precursor cells by stereotaxic intra-striatal injection.

ELIGIBILITY:
Inclusion Criteria:

1. Primary Parkinson's disease patients，a history over 5 years，females or males;
2. Cannot effectively control the PD or tolerate the side effects of drugs;
3. Hoehn and Yahr Stage 3 or 4 in the off state at screening
4. Age between 50 and 80 years;
5. Dopamine is effective or once;
6. Sign the informed consent

Exclusion Criteria:

1. Atypical Parkinsonian syndrome or only having tremor syndrome;
2. Having been done pallidotomy, DBS, striatum or extrapyramidal surgery;
3. Subjects are using apomorphine or anticoagulant;
4. Subjects used immunosuppressant or antipsychotic drugs in last 3 months;
5. Subjects used botulinum toxin, phenol, or other drugs for the treatment of dystonia or muscle cramps in last 6 months;
6. During the period of active epilepsy preventing epilepsy with antiepileptic;
7. Coagulant function abnormality or other obviously abnormal laboratory test results;
8. Having skin basal cell carcinoma or cervical cancer and other pre-cancerous lesions;
9. Subject has a history of chronic alcohol or drug abuse ;
10. Pregnancy or lactation;
11. Subjects participated in other clinical trials in recent 3 months;
12. Subject is considered as dementia, a serious mental disorder (depression or mania), and personality or behavioral disorders through cognitive and behavioral test;
13. Cannot cooperate on the research;
14. Severe brain atrophy, or existing brain injury such as cerebral infarction, cerebral vascular malformation or trauma;
15. Severe systemic diseases;
16. Severe dyskinesia or frequent "OFF" or "ON" states
17. Severe infectious diseases (eg HIV, HCV, HBV, syphilis positive)
18. Not suitable to participate in this clinical trial assessed by other physicians

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), severe TEAEs as assessed by head MRI and blood examination | 6 months
  Number of subjects with adverse events such as the evidence of graft failure or rejection

SECONDARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) score from baseline | Baseline and 12 months
  The total Unified Parkinson's Disease Rating Scale (UPDRS) score is derived from Part I (Mentation, Behavior and Mood), Part II (Activities of Daily Living) and Part III (Motor Examination). Part I assesses 4 functions; Part II assesses 13 activities of daily living; Part III assesses 14 motor symptoms. Each item is rated on a scale from 0 (normal) to 4 (severe). The minimum total score possible is 0 and the maximum total score possible is 176. Each subject was independently rated by two observers at each study visit and a mean score was calculated for analysis.
Change in DATscan from baseline | Baseline and 12 months
  DATscan is an imaging technology that uses small amounts of a radioactive drug to help determine how much dopamine is available in a person's brain.Its principle is based on using of radiopharmaceutical, which bind to dopamine transporters (DAT).
Change in Hoehn and Yahr Stage from baseline | Baseline and 12 months
  The Hoehn and Yahr scale is a commonly used system for describing how the symptoms of Parkinson's disease progress mainly by observing balance and walk.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Qi, Doctor, Principal Investigator — Institute of Zoology, Chinese Academy of Sciences
Locations (1):
- The first affiliated hospital of Zhengzhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang YK, Zhu WW, Wu MH, Wu YH, Liu ZX, Liang LM, Sheng C, Hao J, Wang L, Li W, Zhou Q, Hu BY. Human Clinical-Grade Parthenogenetic ESC-Derived Dopaminergic Neurons Recover Locomotive Defects of Nonhuman Primate Models of Parkinson's Disease. Stem Cell Reports. 2018 Jul 10;11(1):171-182. doi: 10.1016/j.stemcr.2018.05.010. Epub 2018 Jun 14. PMID 29910127